CLINICAL TRIAL: NCT01866553
Title: A Phase II, Single Arm, Multicenter Study of Nilotinib in Combination With Pegylated Interferon-α2b in Patients With Suboptimal Molecular Response or Stable Detectable Molecular Residual Disease After at Least Two Years of Imatinib Treatment (NordDutchCML009)
Brief Title: Nilotinib Plus Pegylated Interferon-α2b in CML
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: insufficient enrollment
Sponsor: Amsterdam UMC, location VUmc (Other)
Collaborators: Uppsala University Hospital (Other); Novartis (Industry); Merck Sharp & Dohme LLC (Industry)
Responsible Party: Principal Investigator, J.J.W.M. Janssen, MD, PhD, Amsterdam UMC, location VUmc
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NordDutchCML009; 2012-004321-25 (EudraCT Number); NTR 3732 (Other: NTR)
Record Dates: First submitted 2013-05-28; First posted 2013-05-31 (Estimated); Last update posted 2018-10-12 (Actual); Status verified 2018-10

CONDITIONS: Chronic Myeloid Leukemia
Keywords: CML; suboptimal molecular response; nilotinib; pegylated interferon α2b
MeSH Terms: conditions — Leukemia, Myelogenous, Chronic, BCR-ABL Positive | interventions — nilotinib; peginterferon alfa-2b

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Nilotinib, Pegylated interferon α2b (Experimental): Patients will be treated with nilotinib 300 mg BID during the first 3 months. Then the "combination phase" ensues with continued daily nilotinib 300 mg BID combined with PegIFN 25 ug/week for 3 months up to the Month 6 time point. If the patient has no more than grade 1 non-hematological toxicity or grade 2 hematological toxicity, the dose will be increased to 40 μg/w until Month 12. The "follow-up phase" with daily nilotinib 300 mg BID covers the next 12 months period (Month 12 to 24). until Month 12, which is followed by monotherapy phase of nilotinib 300 mg BID. Overall study duration for the individual patient is 24 months.
  Interventions: Drug: Nilotinib; Drug: Pegylated interferon α-2b

INTERVENTIONS:
Drug: Nilotinib — 300 mg capsule BID oral use
  Other Names: Tasigna
Drug: Pegylated interferon α-2b — 25 - 40 microgram per week for subcutaneous use
  Other Names: PegIFN; PegIntron; Pegylated interferon alfa-2b; Peginterferon alfa-2b

SUMMARY:
The purpose of this trial is to assess the effect of switching CML patients, who have been treated with imatinib ≥ 2 years and who have stable detectable molecular residual disease between 0.01-1.0% (IS), to the combination of Nilotinib and PegIFN, in terms of the proportion of patients who achieve confirmed MR4.0.

DETAILED DESCRIPTION:
Study phase: Phase II.

Patient population:

Patients with suboptimal molecular response or stable detectable molecular residual disease after ≥ 2 years of treatment with imatinib (i.e. BCR ABL level between 0.01% and 1% IS).

Study objective:

To assess the effect of switching CML patients, who have been treated with imatinib ≥ 2 years and who have stable detectable molecular residual disease between 0.01-1.0% (IS), to the combination of Nilotinib and PegIFN, in terms of the proportion of patients who achieve confirmed MR4.0.

Study design:

Single arm, open label, multicenter study to assess the efficacy, safety and tolerability of nilotinib 300 mg BID, alone and in combination with PegIFN 25 - 40 μg/week in patients not in CMR. Patients will be treated with nilotinib 300 mg BID at the beginning of the study to establish the tolerability before adding PegIFN. Combination treatment will be continued until Month 12, which is followed by monotherapy phase of nilotinib 300 mg BID. Overall study duration for the individual patient is 24 months.

ELIGIBILITY:
Inclusion Criteria:

1. Patients ≥ 18 years
2. At diagnosis CML in chronic phase
3. Documented complete cytogenetic response by bone marrow (standard cytogenetics) or peripheral blood BCR ABL <1% IS
4. Persistent disease demonstrated by two PCR positive tests (i.e. BCR ABL level between 0.01% and 1% IS) which have been performed during the past 9 months and more than 10 weeks apart. One of these should be performed within 1 month of registration
5. Treatment with imatinib for at least 2 years with 400 mg and at a stable dose (i.e. the dose has not changed in the previous 6 months)
6. No other current or planned anti leukemia therapies
7. ECOG Performance status 0,1, or 2
8. Adequate organ function as defined by:

   1. Total bilirubin <1.5 x ULN. Does not apply to patients with isolated hyperbilirubinemia (e.g. Gilbert's disease) grade <3.
   2. ASAT and ALAT <2.5 x ULN.
   3. Serum amylase and lipase ≤1.5 x ULN.
   4. Alkaline phosphatase ≤2.5 x ULN.
   5. Creatinine clearance >30 ml/min.
   6. Mg++, K+ ≥LLN.
9. Life expectancy > 12 months in the absence of any intervention
10. Patient has given written informed consent

Exclusion Criteria:

1. Prior accelerated phase or blast crisis.
2. Patient has received another investigational agent within last 6 months.
3. Previous treatment with nilotinib or dasatinib.
4. Prior stem cell transplantation.
5. Impaired cardiac function including any one of the following:

   1. Inability to monitor the QT/QTc interval on ECG.
   2. Long QT syndrome or a known family history of long QT syndrome.
   3. Clinically significant resting brachycardia (<50 bpm).
   4. QTc >450 msec on baseline ECG (using the QTcF formula). If QTcF >450 msec and electrolytes are not within normal ranges, electrolytes should be corrected and then the patient re screened for QTc.
   5. Myocardial infarction within 12 months prior to starting study.
   6. Other clinically significant uncontrolled heart disease (e.g. unstable angina, congestive heart failure or uncontrolled hypertension).
   7. History of or presence of clinically significant ventricular or atrial tachyarrhythmias.
6. Known atypical BCR ABL transcript not quantifiable by standard RQ PCR
7. History of active malignancy during the past 5 years with the exception of basal carcinoma of the skin or carcinoma in situ of cervix uteri or breast.
8. Acute liver disease or cirrhosis.
9. Previous or active acute or chronic pancreatic disease.
10. Another severe and/or life threatening medical disease.
11. History of significant congenital or acquired bleeding disorder unrelated to cancer.
12. Impairment of gastrointestinal (GI) function or GI disease that may significantly alter the absorption of study drug.
13. Patients actively receiving therapy with strong CYP3A4 inhibitors and the treatment cannot be either discontinued or switched to a different medication prior to starting study drug.
14. Patients who are currently receiving treatment with any medications that have the potential to prolong the QT interval and the treatment cannot be either discontinued or switched to a different medication prior to starting study drug.
15. Patients who are pregnant, breast feeding, of childbearing potential without a negative pregnancy test prior to baseline; male or female of childbearing potential unwilling to use contraceptive precautions throughout the trial (post menopausal women must be amenorrheic for at least 12 months to be considered of non childbearing potential).
16. Interruption of imatinib therapy for a cumulative period in excess of 21 days in the preceding 3 months.
17. Major toxicity on imatinib in past 3 months.
18. History of non compliance, or other inability to grant informed consent.
19. Past or present history of alcohol abuse, use of illicit drugs, or severe psychiatric disorders, including depression.
20. Known hypersensitivity to any interferon preparation.
21. Autoimmune hepatitis or a history of autoimmune disease.
22. Pre existing thyroid disease unless it can be controlled with conventional treatment.
23. Epilepsy and/or compromised central nervous system (CNS)function.
24. HCV/HIV patients.
25. Poorly controlled diabetes mellitus(i.e. HbA1c >9.0) or clinically relevant diabetic complications such as neuropathy, retinopathy, nephropathy, coronary or peripheral vascular disease.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2013-04 (Actual); Primary Completion 2016-04-08 (Actual); Study Completion 2016-05-01 (Actual)

PRIMARY OUTCOMES:
the proportion of patients achieving confirmed MR4.0. | 12 months
  An interim efficacy analysis will be prepared after 40 patients have completed 12 months study treatment.If already a sufficient number of patients have achieved the efficacy endpoint i.e. a 25% increase in MR4.0 rate (from 48% in ENEStcmr to 73% in this study). Using Fleming's method, we have indication of superior efficacy of the combination if 29 or more patients achieve MR4.0, and thereafter may stop inclusion in the study.

SECONDARY OUTCOMES:
the number of patients experiencing grade 3 or more adverse events | 6 months
  A safety interim analysis by a Safety Monitoring Committee (SMC) is planned after 15 patients have completed the Month 6 study assessment, i.e. after 3 months of the combination therapy. The study should be stopped if 4 out of 5, 6 out of 10 or 8 out of 15 patients experience grade 4 hematological toxicity, or grade 3 non hematological toxicity after 3 months of PegIFN treatment.
The proportion of patients who complete the planned 9 months of combination therapy with PegIFN (i.e. to Month 12 assessment). | 12 months
  An evaluation of the dose increase from 25 to 40 μg/week will be performed when 15 patients have passed the 9 month time point (i.e 3 months on 40 μg/week).

OTHER OUTCOMES:
Disease progression | 24 months
Overall Survival | 24 months
Quality of Life | 24 months
the adherence to combination treatment | 24 months
the percentage of patients who lose response after cessation of IFN between Month 12 and 18 | 24 months

CONTACTS AND LOCATIONS:
Overall Officials: Jeroen Janssen, MD, PhD, Principal Investigator — Amsterdam UMC, location VUmc
Locations (5):
- Aarhus University Hospital, Aarhus, Denmark
- Helsinki University Hospital, Helsinki, Finland
- VU University Medical Center, Amsterdam, Netherlands
- Trondheim University Hospital, Trondheim, Norway
- Uppsala University Hospital, Uppsala, Sweden

REFERENCES:
- [Derived] Geelen IGP, Gullaksen SE, Ilander MM, Olssen-Stromberg U, Mustjoki S, Richter J, Blijlevens NMA, Smit WM, Gjertsen BT, Gedde-Dahl T, Markevarn B, Koppes MMA, Westerweel PE, Hjorth-Hansen H, Janssen JJWM. Switching from imatinib to nilotinib plus pegylated interferon-alpha2b in chronic phase CML failing to achieve deep molecular response: clinical and immunological effects. Ann Hematol. 2023 Jun;102(6):1395-1408. doi: 10.1007/s00277-023-05199-1. Epub 2023 Apr 29. PMID 37119314